CLINICAL TRIAL: NCT04104815
Title: A Study to Evaluate the GI Tolerance and Acceptability of a New Thickener for Dysphagia Patients
Brief Title: GI Tolerance and Acceptability of a New Thickener
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Timing
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DA26
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Gastro-intestinal Tolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Thickener (Experimental): Powder thickener
  Interventions: Other: Experimental Thickener

INTERVENTIONS:
Other: Experimental Thickener — Use to thicken liquids

SUMMARY:
The current study is designed to evaluate the gastrointestinal tolerance and acceptability of a new thickener for dysphagia patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an ICF approved by an IRB/IEC, and provided applicable privacy authorization prior to any participation in the study.
* Subject is diagnosed with dysphagia.
* Subject is under the care of a Speech and Language Therapist and is currently using a thickener.
* Subject currently has normal GI function.
* Subject is interested in participating in the study, willing to comply with the study protocol and product.
* Subject who is able to consent and is able to evaluate the product.

Exclusion Criteria:

* Subject has a normal swallow.
* Subject at high risk of aspiration with oral fluids requiring nil by mouth and enteral tube feeding.
* Subject has impaired renal function.
* Subject has liver failure, decompensated chronic liver disease, active hepatitis B or C receiving treatment, or hepatic encephalopathy.
* Subject has severe dementia or unable to communicate or consent or delirium, eating disorder, history of significant neurological or psychiatric disorder affecting abilities to answer questions, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures.
* Participant is known to be allergic or intolerant to any ingredient found in the study product.
* Participation in another study that has not been approved as a concomitant study.
* Subject has a clinical condition that is contraindicated with this product such as hepatic and renal disease.
* Subject has a clinical condition which may interfere with gastrointestinal tolerance.
* Subject is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Bristol Stool Scale | Study Day 1 to Study Day 7
  The Bristol Stool Scale is used to describe the consistency of stools. Numbers 1-7 are assigned to stools based on descriptions on the scale from hard to liquid.
HCP Product Satisfaction Questionnaire | Study Day 7
  5 Questions; 3 of the questions utilize a 5 point scale in the positive direction; 2 of the questions are closed categories yes or no.
Palatability of Study Product | Study Day 1 and Study Day 7
  A 5 point scale in the positive direction
Product Compliance | Study Day 1 to Study Day 7
  Patient thickened fluids consumption records

OTHER OUTCOMES:
Weight | Study Day 1 and Study Day 7
  Weight in Kg
Medications | Study Day 1 to Study Day 7
  Current medication use
Thickness of drinks prescribed | Study Day 1 to Study Day 7
  Current prescription per IDDSI guidelines
Medical aetiology of dysphagia | Study Day 1 and Study Day 7
  Current documentation of medical aetiology

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stevenson, Study Chair — Abbott Nutrition

IPD SHARING:
Plan to Share IPD: No